CLINICAL TRIAL: NCT06327087
Title: Appetite and Energy Balance Parameters Across the Menstrual Cycle
Brief Title: Appetite and Dietary Intake Across the Menstrual Cycle
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Sarah Purcell, Assistant Professor, University of British Columbia
Other Study IDs: 22-00874
Record Dates: First submitted 2024-02-27; First posted 2024-03-25 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Appetitive Behavior; Healthy; Dietary Habits
Keywords: energy expenditure; appetite sensations; diet
MeSH Terms: conditions — Appetitive Behavior; Feeding Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — Observational study in the late follicular and mid-luteal phase

SUMMARY:
Lay language summary: Women are younger and menstruating about monthly ("pre-menopausal") often have fluctuations in the food they eat ("dietary intake") across the menstrual cycle. However, relationships between food intake and appetite, metabolism, body composition (i.e., the proportion of muscle and fat), physical activity and premenstrual symptoms have not been reported. This study will measure appetite and food intake in laboratory and usual life settings in healthy pre-menopausal women in two hormonally different parts of the menstrual cycle. Data on ovarian hormones, metabolism, body composition, physical activity and premenstrual symptoms will also be collected to assess their potential relationship with food intake.

DETAILED DESCRIPTION:
Energy balance parameters (dietary intake and energy expenditure) are influenced by gonadal hormones, such as estradiol and progesterone that fluctuate across the menstrual cycle in pre-menopausal women. Dietary intake varies across the menstrual cycle, with higher self-reported energy intake in the luteal phase. However, it is unclear how physiological and behavioral parameters such as appetite, resting metabolic rate, body composition, physical activity, or premenstrual symptoms relate to energy intake fluctuations. Furthermore, only two studies have measured free-living objective dietary intake across the menstrual cycle, neither of which have measured other aspects of energy balance in detail. This study will help address these knowledge gaps by characterizing several aspects of energy balance in both laboratory and free-living settings in healthy pre-menstrual women across the menstrual cycle. Twenty-three women (for complete data on n=18) aged 18-35 without major comorbidities and with normal menstrual cycles will be enrolled in an observational trial. In addition to a baseline visit to measure body composition, participants will undergo two 4.5-hour study visits, one of which will occur in the follicular phase and the other in the luteal phase (as confirmed with multiple low-burden methods including self-reported menstrual cycle history and urinary luteinizing hormone). Participants will be given a two-day run-in diet prior to each study day to ensure energy balance. On each study day visit, participants will undergo a resting metabolic rate test followed by a series of fasting saliva samples quantitatively pooled to measure estradiol and progesterone. Following collection of fasted ratings of appetite, participants will be provided with a standard breakfast meal. Appetite ratings will be repeated 30, 60, 90, 120, 150, and 180 minutes after the meal. Questionnaires related to eating behavior will also be completed during this time. After the 180-minute timepoint, participants will be provided with a buffet-like lunch meal with instructions to eat as much or as little as they would like; this will allow measurement of ad libitum dietary intake at a single meal. To assess free-living ad libitum dietary intake, participants will receive three days of food boxes tailored to their preferences, with uneaten food returned at the end of the three-day period. After each study visit, participants will be asked to record their dietary intake and appetite (three days) and wear and activity monitor (seven days). Differences in outcomes between visits will be assessed using paired samples t-tests and relationships among variables will be assessed via Pearson correlations. This study will provide preliminary evidence of the factors associated with dietary intake fluctuations across the menstrual cycle and provide essential preliminary data that could inform future weight management and health-promotion strategies.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age: 18 - 35 years
* Nulliparous
* Body mass index (BMI): 18.5 - 24.9 kg/m2
* Premenopausal, with regular menstrual cycle (every 21-38 days, by self-report)
* Sedentary or recreationally active, defined as: <300 minutes per week of voluntary exercise at moderate intensity or greater over the past 12 weeks
* Not currently pregnant or lactating, not planning to become pregnant in the next 12 weeks
* Ability and willingness to fast for 12 hours before each study day visit
* If applicable:

  * For people who occasionally (i.e., <1x/day) use cannabis (including cannabidiol-based products): ability and willingness to abstain from cannabis for two days prior to each study day visit, the day of each study visit, and during each ad libitum diet phase.
  * For people who use cannabis daily: ability and willingness to continue to use the exact same amount of cannabis as they normally use for two days prior to each study day visit, the day of each study visit, and during each ad libitum diet phase.

Exclusion Criteria:

* Current or previous major comorbidities, by self-report, including:

  * Cardiovascular diseases
  * Diabetes (type 1 or type 2)
  * Cancer
  * Thyroid diseases
  * Human immunodeficiency virus or hepatitis B or C
  * Renal diseases
  * Hepatic diseases
  * Polycystic ovary syndrome
* Uncontrolled/untreated (self-report):

  * Hypertension (or measured diastolic blood pressure > 100 mm HG or systolic blood pressure > 160 mm HG)
  * Dyslipidemia
  * Sleep disorders
  * Any other condition that may affect appetite and energy balance
* Currently or in the past six months:

  * Use of oral contraceptive pills, or any other hormone-related birth control
  * Progestin-releasing intrauterine device
  * Use of any hormone therapy/medication ( except medication for thyroid conditions, that has not been altered for >6 months)
  * Use of regular medication that may affect appetite, energy balance, or sleep
  * Regular use of tobacco or nicotine products
* Starting any new prescription medication within two weeks of the first study day visit or during the study
* If applicable, inability to abstain from supplements or herbal products that may impact sex hormones (e.g., chastetree, phytoestrogens, calcium d glucarate, soy isoflavones, maca, black cohosh, red raspberry, etc.) for two weeks prior to the first study day visit and until the second study day visit and free-living assessments are completed.
* Working night shifts or traveling across more than 2 time zones within two weeks of and throughout the study
* Food intolerances or allergies that cannot be accommodated
* History of surgical procedure for weight loss at any time (e.g. gastroplasty, gastric bypass, gastrectomy or partial gastrectomy, adjustable banding, gastric sleeve); history of extensive bowel resection for other reasons
* Current alcohol or substance abuse (score >1 on the cut down-annoyed-guilty-eye opener [CAGE] questionnaire)
* Current or past history of eating disorders including anorexia nervosa, bulimia, binge eating disorder (self-report or score >20 on the Eating Attitudes Test - 26 [EATS-26] questionnaire)
* Current severe depression or history of severe depression within the previous year, based on score > 30 on Beck Depression Inventory (BDI)
* Weight loss >5kg in past 12 weeks for any reason
* Weight loss of >20 kgs in past 3 years for any reason

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: Healthy sedentary or recreationally active females with normal menstrual cycles
Sampling Method: Non-Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Energy intake | 1 hour
  Ad libitum intake at lunch; difference between energy in weighed food before and after consumption in a laboratory setting
Hunger area under the curve | 3 hours (pre and 30, 60, 90, 120, 150, and 180 minutes after breakfast)
  Repeated visual analog scale (0-100mm) ratings of hunger after a standard breakfast meal
Satiety area under the curve | 3 hours (pre and 30, 60, 90, 120, 150, and 180 minutes after breakfast)
  Repeated visual analog scale (0-100mm) ratings of satiety after a standard breakfast meal
Prospective food consumption area under the curve | 3 hours (pre and 30, 60, 90, 120, 150, and 180 minutes after breakfast)
  Repeated visual analog scale (0-100mm) ratings of prospective food consumption after a standard breakfast meal

SECONDARY OUTCOMES:
Free-living ad libitum energy intake | 2.5 days following study visit
  Ad libitum intake; difference between energy in weighed food before and after consumption, provided to participants in free-living environments
Resting metabolic rate | 30 minutes
  Resting metabolic rate, via indirect calorimetry (metabolic cart)
Body composition | 30 minutes
  Fat mass and fat-free mass from dual X-ray absorptiometry
Estradiol | 5 minutes
  Concentration of circulating estradiol, measured from saliva
Progesterone | 5 minutes
  Concentration of circulating progesterone, measured from saliva
Physical activity patterns | 7 days
  Physical activity patterns (e.g., steps/day, time spent sitting, or in moderate-to-vigorous physical activity) from activPAL accelerometers

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia - Okanagan, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
De-identified data will be made available to researchers upon reasonable request.